CLINICAL TRIAL: NCT02842801
Title: Hip Manipulation in Young Adults With Complaints of Pain in the Groin, Lateral Hip or Buttock: Which Patients Will Have an Immediate Benefit?
Brief Title: Hip Manipulation in Young Adults With Groin, Lateral Hip or Buttock Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Sharon Wang-Price, Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18174
Record Dates: First submitted 2016-07-20; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Hip Strain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hip Manipulation (Other): Hip manipulation: high velocity low amplitude thrust mobilization
  Interventions: Other: Hip manipulation

INTERVENTIONS:
Other: Hip manipulation — High-amplitude and low-velocity thrust mobilization

SUMMARY:
The purpose of the study is to identify the characteristics of young adults with pain in the groin, lateral hip or buttock who will benefit from manipulation of the hip.

DETAILED DESCRIPTION:
Unlike older adults with hip osteoarthritis, young adults with pain in the groin, lateral hip or buttock do not have general loss of ROM, but have a specific directional motion loss, such as hip flexion and internal rotation. Therefore, the most common manual therapy designed to gradually improve hip range of motions (ROM) for osteoarthritis, long axis distraction, may not be appropriate for treating young adults with hip pain. A manipulation technique, unrestrained femoral internal rotation (UFIR), was designed specifically for treating young adults' hip pain. Manipulation is a procedure that involves the use of a high- amplitude and low-velocity thrust at the mid or end range of a restricted joint for the purpose of improving range of motion (ROM) within the joint and the ability of the joint to tolerate loads.

Although clinicians routinely use this hip manipulation technique for treating young adults' hip pain with satisfying success, no study yet has been conducted to examine the effectiveness of this hip manipulation technique. The investigators are interested in identifying which young adults with pain in the groin, lateral hip or buttock would benefit from this hip manipulation.

Adverse effects of this manipulation have been reported to be none to mild. Mild soreness or muscle tenderness at the posterior greater trochanter region has been reported. In a preliminary study on the UFIR manipulation of 35 participants, 5 reported mild discomfort immediately after manipulation, but no participants reported adverse effects of a UFIR manipulation.

Purpose of the Study:

The purpose of the proposed study is to identify the characteristics of young adults with pain in the groin, lateral hip or buttock who will benefit from manipulation of the hip.

Research question:

What are the predictors for a positive outcome of hip manipulation on young adults with groin, lateral hip or buttock pain?

Procedures:

At the beginning of the study, all participants with groin/lateral hip/buttock pain will be informed of the risks, benefits and procedures of the study. Once the participants agree to participate, they will be asked to sign a written consent form approved by the TWU Institutional Review Board - Dallas. Once each participant signs the consent form, a number will be assigned to the participant and all forms to be used will be marked with this number. All data collection including the testing and treatment will be performed at the Texas Woman's University (TWU) - Dallas, Lab #8113, or in a private treatment room at the Physical Therapy & Injury Specialist clinic, Englewood, CO. Each participant will come twice with 24-48 hours between visits.

1st Visit: On the first visit, all participants will be asked to fill out an intake form and a medical questionnaire to further determine the eligibility of each participant. Next, one of the investigators will perform a neurological exam, including dural tests, femoral nerve tests, deep tendon reflexes, key muscle tests and Babinski/Hoffman to rule out lumbar or neurologic involvement. If a participant is found to have a positive neurological test, the participant will be excluded from the study.

Outcome Measures and Special Questions:

Once the participant is determined to be eligible for the study, each participant will be asked to complete the following 4 questionnaires:

1. Numerical Pain Rating Scale (NPRS) with body charts
2. Lower Extremity Functional Scale
3. The Copenhagen Hip and Groin Outcome Score (HAGOS)
4. Special questions for functional activities.

The reliability and validity of the NPRS, LEFS and HAGOs have been shown to be reliable and valid. The special questions were used to describe the characteristics of the participants who are young adults with groin, lateral hip or buttock pain.

Physical Examination

A standard physical therapy examination specific to the hip will be performed by the investigator who will not perform the hip manipulation:

1. Functional tests: 3 functional tests will be assessed: deep squat, hurdle and inline lunge.
2. Palpation tests: 11 palpation tests will be examined. The surrounding bony landmark and soft tissue also will be palpated for tenderness and abnormality. To improve test accuracy, the investigators will video tape 2 palpation tests: single leg stand and single leg stance.
3. Range of motion (ROM) measurements: 8 hip ROMs will be measured in supine and prone. A universal goniometer will be used to take all of hip ROMs. Two measurements will be taken for each motion, and the average of the two will be used for data analysis.
4. Manual muscle strength tests: 8 hip manual muscle tests will be performed in sitting, supine, sidelying and prone positions:

   * Sitting: flexion
   * Supine: flexion, internal rotation and external rotation
   * Sidelying: abduction
   * Prone: extension, internal rotation and internal rotation
5. Provocation tests of lumbar, sacroiliac and hip joints.

Intervention:

The other investigator, a licensed physical therapist and different from the one who performed physical examination as described above, will perform the intervention technique, hip manipulation UFIR. During the manipulation, the participant will be asked to lie on the unaffected side with the affected side up, their hip(s) flexed to approximately 30 degrees, and knees flexed to approximately 50-70 degrees. Pillows will be place between the participant's knees as needed for comfort. The investigator will stabilize the anterior inferior iliac spine (ASIS) and ilium with the fingers of one hand and place the thumb on the posterior aspect of the greater trochanter of the involved hip. The participant will be asked for verbal approval prior to receiving the manipulation. The manipulation will be performed with the investigator's non-stabilizing hand, by thrusting the greater trochanter anteriorly with an internal rotation moment.

The manipulation will be performed on the involved side. If the participant or the investigator feels a cavitation or shift in the hip joint after the first manipulation, the intervention will be considered complete. If no cavitation/shift is heard or felt by the participant or the investigator after the first manipulation, the investigator will repeat the manipulation up to a maximum of three times. The manipulation will be performed by either of two physical therapists who have specialized in manual therapy, and have been certified after participating in an extensive clinical education and examination process.

Post Intervention After the hip manipulation intervention, the investigator will advise the participant to continue any regular activity but to not perform new activities. In addition, the participant will be asked to fill out the NPRS with body charts (Appendix E) and the Global Rating of Change (GROC) Scale (Appendix M).16 The participant will reminded of the second visit day and appointment time within 24-48 hours.

2nd Visit During the 2nd visit, the same investigator who has evaluated the participant on his/her 1st visit will perform the same physical exam as described on the first visit, with the same measurement or reporting details. Following this physical exam, the participant will be asked to fill out the NPRS with body charts, LEFS, HAGOS and GROC forms. There will be no further treatment for the purpose of the study.

Data Analysis The participants will be dichotomized into two groups based on their response to the hip manipulation: successful or non-successful. Success will be defined as 2 points or greater change in the NPRS or 4 points or greater change in the GROC. These criteria will be used as reference standards to dichotomize the participants for all variables collected from patient's history, self-reported questionnaires and physical exam. Regression analysis will be used to examine significant predictors/characteristics for a successful outcome of hip manipulation on young adults with groin, lateral hip or buttock pain.

ELIGIBILITY:
Inclusion Criteria:

* The eligible participants will be young adults of both genders between the ages of 18-40 who have complaints of groin, lateral hip and/or buttock pain.

Exclusion Criteria:

* Participants will be excluded from participating in this study if they have any of the following medical or surgical history. These factors may affect the results of the study:

  1. Impaired general health, e.g. fibromyalgia, chronic fatigue syndrome, cancer etc.
  2. Neurologic or neurovascular dysfunction
  3. History of peripheral vascular disease, diabetes or abdominal aneurysm
  4. History of hip joint pathology, such as slipped epiphysis, Legg Calve Perthes, significant congenital hip dysplasia, and hip dislocation,
  5. History of systemic disease affecting the musculoskeletal or neuromuscular systems, including inflammatory arthritides, connective tissue diseases, multiple sclerosis, muscular dystrophy, and cerebral vascular diseases
  6. Known instabilities of hip or sacroiliac joint
  7. History of low back and lower extremity surgery, e.g. total hip replacement, total knee replacement, lumbar laminectomy.
  8. A diagnosed hip labral tests or clicking, catching, popping or hypermobility signs with hip labral tear tests
  9. Amputee of lower extremity
  10. Fracture hip or spine
  11. Infection in spine or lower extremities
  12. Hip ROM loss in all directions
  13. Pregnant or up to 12 weeks post-partum
  14. Bleeding or clotting disorders
  15. Osteoporosis
  16. Treated with hip manipulation in past 12 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Global Rating of Change (GROC) Scale | Short-term
  24-48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wang-Price, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No